CLINICAL TRIAL: NCT01866189
Title: Assessment of Hypoxic Tissues in Acute Ischemic Stroke With 18F-FMISOnidazole PET and Comparison With MRI : A Prospective Multicenter Study
Brief Title: Identification of Hypoxic Brain Tissues by F-MISO PET in Acute Ischemic Stroke
Acronym: STROKE F-MISO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: default recruitment
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11 252 01
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; hypoxic tissues; F-MISO uptake; Magnetic Resonance Imaging; F-MISO Positon Emission Tomography
MeSH Terms: conditions — Ischemic Stroke | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy; tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET and MRI (Experimental): Included patients will have F-MISO PET followed by brain MRI (MRI-1)(diffusion, FLAIR, perfusion, TOF) as soon as possible after stroke onset (less than 36 hours). A second brain MRI (MRI-2) will be performed on day 7.
  Interventions: Other: PET and MRI

INTERVENTIONS:
Other: PET and MRI — F-MISO PET followed by brain MRI (MRI-1)(diffusion, FLAIR, perfusion, TOF)
  Other Names: TEP

SUMMARY:
This study is a French multicenter prospective study including 5 stroke units with available MRI and F-MISO PET for patients with acute ischemic stroke.

Background and Purpose: 18F-Fluoromisonidazole (FMISO) PET has been used to identify hypoxic tissues in animals and stroke patients. While MRI has become the gold standard acute stroke imaging, no published study has compared FMISO PET and MRI.

The aim of this prospective study is to identify hypoxic tissues in 40 patients with acute ischemic stroke with F-MISO PET and to compare the location and the outcome of these hypoxic cells with MRI datas (weighted diffusion and FLAIR) and to clinical outcome.

DETAILED DESCRIPTION:
40 prospective patients (aged 18 to 85 years) will be included in the first 36 hours after ischemic stroke onset.

The study period will be 2 years. Included patients will have F-MISO PET followed by brain MRI (MRI-1)(diffusion, FLAIR, perfusion, TOF) as soon as possible after stroke onset (less than 36 hours). A second brain MRI (MRI-2) will be performed on day 7.

The aim of the study is to locate hypoxic tissues and to compare with ischemic tissues defined by diffusion and FLAIR MRI sequences, with MRI evolution, and with clinical status at day 7 and day 90.

Inclusion criterias

* Patients aged 18-85 years with encephalic brain ischemic stroke,
* defined stroke onset,
* NIHSS 5 to 20,
* F-MISO Pet and MRI available <36 hours after stroke onset,

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years with encephalic brain ischemic stroke,
* defined stroke onset,
* NIHSS 5 to 20,
* F-MISO Pet and MRI available <36 hours after stroke onset,
* Written consent signed by patient or family

Exclusion Criteria:

* contraindication to MRI
* comatous status
* 5 < NIHSS > 20
* non ischemic stroke
* brainstem stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
volume and location of F-MISO uptake in stroke patients | acute phase of brain ischemia < 36 hours

SECONDARY OUTCOMES:
comparison of F-MISO uptake areas and ischemic lesions defined by weighted diffusion and FLAIR on | acute phase of brain ischemia < 36 hours